CLINICAL TRIAL: NCT00555815
Title: Intraoperative Hygiene Measures and Rates of Surgical Wound Infection in General Surgery
Brief Title: Intraoperative Hygiene Measures and Surgical Site Infections
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: 1.05.01.30.-17
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Surgery; Surgical Site Infection; Hygiene; Discipline; Colorectal Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Extended hygiene measures
- 2: Standard hygiene measures

SUMMARY:
Surgical site infections are associated with high morbidity and cost Hypothesis: Extended intraoperative hygiene measures decrease surgical site infections in general surgery compared to standard hygiene measures.

DETAILED DESCRIPTION:
Intraoperatively two types of hygiene measures were performed randomly: standard and extensive. Standard hygiene measures included empiric accepted measures (e.g. gloves, masks, disinfection). Extensive hygiene measures included among others: double gloving, astro caps, extensive disinfection, extensive intraoperative rinsing. In addition, intraoperative adherence to the rules of asepsis were registered by an independent observer.

Patients were followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing surgical operation in one of two assigned operative theaters. Only initial operations are studied

Exclusion Criteria:

* Previous inclusion into study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients undergoing general surgery in university hospital
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2005-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Surgical site infection 30 days postoperative | 30 days

SECONDARY OUTCOMES:
Adherence to rules of asepsis by members of the surgical team | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Candinas, MD, Study Director — Department of Visceral and Transplant Surgery
Locations (1):
- Department of Visceral and Transplant Surgery, University hospital, Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Beldi G, Bisch-Knaden S, Banz V, Muhlemann K, Candinas D. Impact of intraoperative behavior on surgical site infections. Am J Surg. 2009 Aug;198(2):157-62. doi: 10.1016/j.amjsurg.2008.09.023. Epub 2009 Mar 12. PMID 19285307